CLINICAL TRIAL: NCT03170388
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Vehicle Controlled, Parallel-Group, Clinical Study Comparing the Efficacy and Safety of IDP-126 Gel in the Treatment of Acne Vulgaris
Brief Title: A Phase 2, Multicenter, Randomized, Double-Blind, Vehicle Controlled, Parallel-Group, Clinical Study in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V01-126A-201
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Results first posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized, Double-Blind, Vehicle Controlled, Parallel-Group
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- IDP-126 Gel (Experimental): Gel
  Interventions: Drug: IDP-126 Gel
- IDP-126 Component A (Active Comparator): Component A
  Interventions: Drug: IDP-126 Component A
- IDP-126 Component B (Active Comparator): Component B
  Interventions: Drug: IDP-126 Component B
- IDP-126 Component C (Active Comparator): Component C
  Interventions: Drug: IDP-126 Component C
- IDP-126 Vehicle Gel (Placebo Comparator): Vehicle Gel
  Interventions: Drug: IDP-126 Vehicle Gel

INTERVENTIONS:
Drug: IDP-126 Gel — Gel
  Arms: IDP-126 Gel
Drug: IDP-126 Component A — Component A
  Arms: IDP-126 Component A
Drug: IDP-126 Component B — Component B
  Arms: IDP-126 Component B
Drug: IDP-126 Component C — Component C
  Arms: IDP-126 Component C
Drug: IDP-126 Vehicle Gel — Vehicle Gel
  Arms: IDP-126 Vehicle Gel

SUMMARY:
A Phase 2, Multicenter, Randomized, Double-Blind, Vehicle Controlled, Parallel-Group, Clinical Study in the Treatment of Acne Vulgaris

DETAILED DESCRIPTION:
A Phase 2, Multicenter, Randomized, Double-Blind, Vehicle Controlled, Parallel-Group, Clinical Study Comparing the Efficacy and Safety of IDP-126 Gel in the Treatment of Acne Vulgaris

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 9 years of age and older.
2. Written and verbal informed consent must be obtained. Subjects less than age of consent must sign an assent for the study and a parent or a legal guardian must sign the informed consent (if subject reaches age of consent during the study they should be re-consented at the next study visit).
3. Subject must have an EGSS of 3 (moderate) or 4 (severe) at the baseline visit.
4. Subjects with a facial acne inflammatory lesion (papules, pustules, and nodules) count no less than 20, but no more than 100.
5. Subjects with a facial acne non-inflammatory lesion (open and closed comedones) count no less than 30, but no more than 150.
6. Subjects with 2 or fewer facial nodules

Exclusion Criteria:

1. Use of an investigational drug or device within 30 days of enrollment or participation in a research study concurrent with this study.
2. Any dermatological conditions on the face that could interfere with clinical evaluations such as acne conglobata, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, gram negative folliculitis, dermatitis, eczema.
3. Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive.
4. Subjects with a facial beard or mustache that could interfere with the study assessments.
5. Subjects with more than 2 facial nodules.
6. Evidence or history of cosmetic-related acne.

Ages: 9 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 741 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Bausch Health Americas, Inc.
Locations (34):
- United States (29):
  - Valeant Site 02, Hot Springs, Arkansas
  - Valeant Site 07, Fremont, California
  - Valeant Site 08, Sacramento, California
  - Valeant Site 09, Denver, Colorado
  - Valeant Site 11, Boynton Beach, Florida
  - Valeant Site 13, North Miami Beach, Florida
  - Valeant Site 12, Sanford, Florida
  - Valeant Site 10, West Palm Beach, Florida
  - Valeant Site 15, Marietta, Georgia
  - Valeant Site 14, Snellville, Georgia
  - Valeant Site 16, Boise, Idaho
  - Valeant Site 17, Overland Park, Kansas
  - Valeant Site 18, Louisville, Kentucky
  - Valeant Site 19, Louisville, Kentucky
  - valeant Site 21, Glenn Dale, Maryland
  - Valeant Site 20, Needham, Massachusetts
  - Valeant Site 22, Detroit, Michigan
  - Valeant Site 24, Morristown, New Jersey
  - Valeant Site 25, Albuquerque, New Mexico
  - Valeant Site 27, New York, New York
  - Valeant Site 26, New York, New York
  - Valeant Site 23, High Point, North Carolina
  - Valeant Site 28, Gresham, Oregon
  - Valeant Site 30, Johnston, Rhode Island
  - Valeant Site 31, Nashville, Tennessee
  - Valeant Site 32, Austin, Texas
  - Valeant Site 33, Pflugerville, Texas
  - valeant Site 34, San Antonio, Texas
  - Valeant Site 35, Norfolk, Virginia
- Canada (5):
  - Valeant Site 01, Winnipeg, Manitoba
  - Valeant Site 05, Barrie, Ontario
  - Valeant Site 06, Oakville, Ontario
  - Valeant Site 04, Peterborough, Ontario
  - Valeant Site 03, Waterloo, Ontario

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gold M, Lain T, Harper JC, Baldwin H, Guenin E, Stein Gold L. Efficacy and Safety of Clindamycin Phosphate 1.2%/Adapalene 0.15%/Benzoyl Peroxide 3.1% Gel: Post Hoc Analysis by Baseline Disease Severity. Dermatol Ther (Heidelb). 2025 Jul;15(7):1867-1882. doi: 10.1007/s13555-025-01440-z. Epub 2025 May 16. PMID 40377868
- [Derived] Stein Gold L, Baldwin H, Kircik LH, Weiss JS, Pariser DM, Callender V, Lain E, Gold M, Beer K, Draelos Z, Sadick N, Pillai R, Bhatt V, Tanghetti EA. Efficacy and Safety of a Fixed-Dose Clindamycin Phosphate 1.2%, Benzoyl Peroxide 3.1%, and Adapalene 0.15% Gel for Moderate-to-Severe Acne: A Randomized Phase II Study of the First Triple-Combination Drug. Am J Clin Dermatol. 2022 Jan;23(1):93-104. doi: 10.1007/s40257-021-00650-3. Epub 2021 Oct 21. PMID 34674160

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IDP-126 Gel | IDP-126 Component A | IDP-126 Component B | IDP-126 Component C | IDP-126 Vehicle Gel
Started | 147 | 150 | 146 | 150 | 148
Completed | 125 | 132 | 133 | 132 | 127
Not Completed | 22 | 18 | 13 | 18 | 21

BASELINE CHARACTERISTICS:
Population: One participant in the IDP-126 Gel group did not receive study medication and thus is not included in the demography population.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDP-126 Gel | IDP-126 Component A | IDP-126 Component B | IDP-126 Component C | IDP-126 Vehicle Gel | Total
Number analyzed (Participants) | 146 | 150 | 146 | 150 | 148 | 740
Age, Continuous [Median (Full Range); unit: years] | 17 [11 to 46] | 17 [10 to 60] | 17 [10 to 45] | 17 [11 to 50] | 17 [11 to 47] | 17 [10 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 86 | 91 | 93 | 89 | 453
  Male | 52 | 64 | 55 | 57 | 59 | 287
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 1 | 2 | 6
  Asian | 10 | 6 | 8 | 9 | 17 | 50
  Native Hawaiian or Other Pacific Islander | 2 | 4 | 0 | 1 | 0 | 7
  Black or African American | 24 | 26 | 30 | 20 | 26 | 126
  White | 98 | 109 | 101 | 109 | 95 | 512
  More than one race | 11 | 4 | 6 | 10 | 8 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Baseline Evaluator's Global Severity Score [Count of Participants; unit: Participants] — The Evaluator's Global Severity Score has grades for acne severity of 0 (Clear), 1 (Almost Clear), 2 (Mild), 3 (Moderate), and 4 (Severe), with higher scores indicating worse severity.
  Participants
    Moderate | 124 | 119 | 124 | 129 | 127 | 623
    Severe | 22 | 31 | 22 | 21 | 21 | 117

OUTCOME MEASURES:

1. Primary Outcome: Inflammatory Lesion Counts
Description: Absolute change from Baseline to Week 12 in mean inflammatory lesion counts
Time Frame: Baseline to Week 12
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Deviation); unit: lesions
Arm/Group | IDP-126 Gel | IDP-126 Component A | IDP-126 Component B | IDP-126 Component C | IDP-126 Vehicle Gel
Number analyzed (Participants) | 146 | 150 | 146 | 150 | 148
lesions | -29.9 (11.86) | -26.7 (11.74) | -24.8 (11.71) | -26.8 (11.69) | -19.6 (12.12)

2. Primary Outcome: Non-inflammatory Lesion Counts
Description: Absolute change from Baseline to Week 12 in mean non-inflammatory lesion counts
Time Frame: Baseline to Week 12
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Deviation); unit: lesions
Arm/Group | IDP-126 Gel | IDP-126 Component A | IDP-126 Component B | IDP-126 Component C | IDP-126 Vehicle Gel
Number analyzed (Participants) | 146 | 150 | 146 | 150 | 148
lesions | -35.5 (16.25) | -29.9 (16.40) | -27.8 (15.97) | -30.0 (16.40) | -21.8 (16.58)

3. Primary Outcome: Percentage of Participants With Success on the Evaluator's Global Severity Score
Description: Success was defined as at least a two grade reduction and clear or almost clear at Week 12. The Evaluator's Global Severity Score has grades for acne severity of 0 (Clear), 1 (Almost Clear), 2 (Mild), 3 (Moderate), and 4 (Severe), with higher scores indicating worse severity.
Time Frame: Baseline to Week 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | IDP-126 Gel | IDP-126 Component A | IDP-126 Component B | IDP-126 Component C | IDP-126 Vehicle Gel
Number analyzed (Participants) | 146 | 150 | 146 | 150 | 148
percentage of participants | 52.5 | 27.8 | 30.5 | 30.3 | 8.1

4. Secondary Outcome: Inflammatory Lesion Count Changes at Week 2, 4, and 8
Description: Absolute change from Baseline to Week 2, 4, and 8 in mean inflammatory lesion counts
Time Frame: Baseline to Week 2, 4, 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | IDP-126 Gel | IDP-126 Component A | IDP-126 Component B | IDP-126 Component C | IDP-126 Vehicle Gel
Number analyzed (Participants) | 146 | 150 | 146 | 150 | 148
lesions
  Week 2 | -14.0 (11.62) | -11.8 (10.80) | -13.8 (10.50) | -13.4 (10.76) | -9.2 (9.58)
  Week 4 | -21.0 (10.33) | -17.1 (12.07) | -18.8 (12.05) | -17.7 (11.49) | -14.8 (10.26)
  Week 8 | -25.8 (11.97) | -23.0 (11.69) | -23.1 (13.95) | -22.8 (9.86) | -17.5 (10.86)

5. Secondary Outcome: Non-inflammatory Lesion Count Changes at Week 2, 4, and 8
Description: Absolute change from Baseline to Week 2, 4, and 8 in mean non-inflammatory lesion counts
Time Frame: Baseline to Week 2, 4, 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | IDP-126 Gel | IDP-126 Component A | IDP-126 Component B | IDP-126 Component C | IDP-126 Vehicle Gel
Number analyzed (Participants) | 146 | 150 | 146 | 150 | 148
lesions
  Week 2 | -12.9 (12.90) | -11.0 (14.31) | -11.2 (10.97) | -11.3 (14.02) | -9.2 (11.94)
  Week 4 | -21.4 (14.33) | -18.6 (13.74) | -15.8 (13.77) | -18.0 (14.35) | -13.7 (11.78)
  Week 8 | -30.5 (15.95) | -25.1 (15.43) | -21.7 (16.08) | -26.8 (14.68) | -17.6 (15.29)

6. Secondary Outcome: Inflammatory Lesion Count Percentage Changes at Week 2, 4, and 8
Description: Percentage change from Baseline to Week 2, 4, and 8 in mean inflammatory lesion counts
Time Frame: Baseline to Week 2, 4, 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | IDP-126 Gel | IDP-126 Component A | IDP-126 Component B | IDP-126 Component C | IDP-126 Vehicle Gel
Number analyzed (Participants) | 146 | 150 | 146 | 150 | 148
percentage change
  Week 2 | -35.89 (29.073) | -30.27 (26.417) | -35.10 (26.442) | -35.23 (26.926) | -24.18 (26.000)
  Week 4 | -54.42 (22.683) | -44.37 (28.511) | -47.55 (28.040) | -46.32 (27.664) | -39.95 (27.304)
  Week 8 | -66.07 (22.239) | -59.07 (25.573) | -59.55 (31.990) | -60.10 (23.863) | -46.61 (27.495)

7. Secondary Outcome: Non-inflammatory Lesion Count Percentage Changes at Week 2, 4, and 8
Description: Percentage change from Baseline to Week 2, 4, and 8 in mean non-inflammatory lesion counts
Time Frame: Baseline to Week 2, 4, 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | IDP-126 Gel | IDP-126 Component A | IDP-126 Component B | IDP-126 Component C | IDP-126 Vehicle Gel
Number analyzed (Participants) | 146 | 150 | 146 | 150 | 148
percentage change
  Week 2 | -27.07 (26.440) | -23.39 (30.433) | -23.72 (22.845) | -24.91 (28.698) | -19.68 (23.194)
  Week 4 | -43.17 (27.162) | -39.28 (26.422) | -33.84 (29.592) | -38.14 (27.765) | -29.53 (26.025)
  Week 8 | -60.05 (25.164) | -52.76 (27.916) | -47.29 (32.982) | -54.17 (26.530) | -37.84 (29.933)

8. Secondary Outcome: Percentage of Participants With Success on the Evaluator's Global Severity Score at Weeks 2, 4, and 8
Description: Success was defined as at least a two grade reduction and clear or almost clear at the visit. The Evaluator's Global Severity Score has grades for acne severity of 0 (Clear), 1 (Almost Clear), 2 (Mild), 3 (Moderate), and 4 (Severe), with higher scores indicating worse severity.
Time Frame: Baseline to Week 2, 4, and 8
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | IDP-126 Gel | IDP-126 Component A | IDP-126 Component B | IDP-126 Component C | IDP-126 Vehicle Gel
Number analyzed (Participants) | 146 | 150 | 146 | 150 | 148
percentage of participants
  Week 2 | 1.49 | 1.35 | 0.71 | 2.68 | 0.00
  Week 4 | 8.17 | 6.77 | 2.79 | 4.27 | 1.36
  Week 8 | 20.46 | 15.97 | 15.26 | 15.75 | 3.51

9. Secondary Outcome: Percentage of Participants With Two Grade Success on the Evaluator's Global Severity Score - at Weeks 2, 4, and 8
Description: Two grade success was defined as at least a two grade reduction. The Evaluator's Global Severity Score has grades for acne severity of 0 (Clear), 1 (Almost Clear), 2 (Mild), 3 (Moderate), and 4 (Severe), with higher scores indicating worse severity.
Time Frame: Baseline to Week 2, 4, and 8
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | IDP-126 Gel | IDP-126 Component A | IDP-126 Component B | IDP-126 Component C | IDP-126 Vehicle Gel
Number analyzed (Participants) | 146 | 150 | 146 | 150 | 148
percentage of participants
  Week 2 | 2.95 | 2.78 | 1.45 | 5.44 | 1.36
  Week 4 | 11.46 | 10.53 | 5.83 | 8.51 | 2.12
  Week 8 | 28.74 | 22.79 | 19.97 | 20.66 | 4.43

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: There were 6 IDP-126, 4 Component A, 2 Component B, 2 Component C, and 2 Vehicle participants excluded from the adverse event analysis since they did not have post-baseline safety evaluations.
Arm/Group | IDP-126 Gel | IDP-126 Component A | IDP-126 Component B | IDP-126 Component C | IDP-126 Vehicle Gel
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/146 | 0/144 | 0/148 | 0/146
Serious Adverse Events (participants affected / at risk) | 1/141 | 0/146 | 0/144 | 3/148 | 0/146
Other Adverse Events (participants affected / at risk) | 30/141 | 29/146 | 6/144 | 19/148 | 7/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-126 Gel (N=141) | IDP-126 Component A (N=146) | IDP-126 Component B (N=144) | IDP-126 Component C (N=148) | IDP-126 Vehicle Gel (N=146)
Sickle cell anemia with crisis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Abortion induced (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-126 Gel (N=141) | IDP-126 Component A (N=146) | IDP-126 Component B (N=144) | IDP-126 Component C (N=148) | IDP-126 Vehicle Gel (N=146)
Application Site Pain (General disorders) | 11 | 16 | 1 | 5 | 1
Application Site Dryness (General disorders) | 9 | 8 | 2 | 9 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 10 | 5 | 3 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact sponsor for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT03170388/Prot_SAP_000.pdf